CLINICAL TRIAL: NCT05485194
Title: Use of a Titanium Bone Screw for Ridge Preservation Following Tooth Extraction
Brief Title: Ridge Preservation Following Tooth Extraction
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No funding was obtained. Therefore, the study never started.
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Se-Lim Oh, Clinical Associate Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: HP-00102697
Record Dates: First submitted 2022-07-31; First posted 2022-08-03 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Alveolar Bone Resorption; Tooth Extraction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Unassisted healing (No Intervention): The extraction sockets in the non-intervention group will be filled with blood clots only.
- Titanium bone screw (TBS) (Experimental): One titanium bone screw (TBS) will be placed over the labial/buccal plate of the extraction socket in the TBS group on the same day of the extraction.
  Interventions: Other: Reducing dimensional changes following tooth extraction
- Alveolar ridge preservation (ARP) (Active Comparator): The extraction socket will be filled with mineralized ground cortical allograft up to the level of the buccal and lingual/palatal bony plates. A resorbable membrane will be trimmed and adapted to cover the grafting material. The flaps will be secured with a monofilament suture.
  Interventions: Other: Reducing dimensional changes following tooth extraction

INTERVENTIONS:
Other: Reducing dimensional changes following tooth extraction — Use of a titanium bone screw for ridge preservation following tooth extraction
  Arms: Alveolar ridge preservation (ARP); Titanium bone screw (TBS)

SUMMARY:
An animal study and our pilot human study demonstrated that placing a smooth-surface titanium bone screw (TBS) over the buccal plate of an extraction socket resulted in less dimensional changes of the alveolar ridge along with no adverse effects. The purpose of this randomized clinical trial is to investigate the effectiveness of TBS application for ridge preservation in comparison to (1) unassisted/non-interventional socket healing and (2) alveolar ridge preservation (ARP) approach using allografts and a membrane.

DETAILED DESCRIPTION:
The participants will be randomized to one of the three groups: the non-intervention, titanium bone screw (TBS), and alveolar ridge preservation (ARP) groups. The sockets in the non-intervention group will be filled with blood clots only. One TBS will be placed over the labial/buccal plate of the extraction socket in the TBS group on the same day of the extraction. Allograft and resorbable collagen membrane will be used for the ARP group.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* a tooth, which is in the area from the central incisor to the second premolar bounded by teeth (or implants) mesiodistally
* a tooth requiring extraction

Exclusion Criteria:

* thyroid dysfunctions
* diabetes mellitus
* history of a chronic use of corticosteroids (>6 months)
* history of oral/intravenous bisphosphonates within the past 2 years
* smoking
* history of other systemic conditions that could affect bone integrity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
The width of the alveolar bone | up to 6 months
  Dimensional changes in the width of the alveolar bone following tooth extraction

CONTACTS AND LOCATIONS:
Overall Officials: Se-Lim Oh, Principal Investigator — University of Maryland School of Dentistry

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shares with other researchers.

REFERENCES:
- [Result] Joseph S, Oh SL, Pae EK, Joshi S. Use of transcortical miniscrews for alveolar ridge preservation following tooth extraction: A pilot study. Clin Oral Implants Res. 2022 Feb;33(2):150-157. doi: 10.1111/clr.13875. Epub 2021 Nov 16. PMID 34741321
- [Result] Melsen B, Huja SS, Chien HH, Dalstra M. Alveolar bone preservation subsequent to miniscrew implant placement in a canine model. Orthod Craniofac Res. 2015 May;18(2):77-85. doi: 10.1111/ocr.12058. Epub 2014 Nov 18. PMID 25403977